CLINICAL TRIAL: NCT05631925
Title: Comparison of Two Different Anesthesia Methods During Oocyte Retrieval for in Vitro Fertilization
Brief Title: Comparison of Two Different Anesthesia Methods in IVF Procedure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Sevgi Bilgen, Associate Professor, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: SBilgen
Record Dates: First submitted 2022-11-02; First posted 2022-11-30 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Oocyte Retrieval

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group bolus (Active Comparator): Propofol will be administered in bolus doses of 0.5mg/kg. Doses will be determined according to the clinical condition of the patient.
  Interventions: Drug: propofol bolus
- Group infusion (Active Comparator): Propofol will be administered as 10mg/kg/hour infusion. The infusion dose will be adjusted so that the Bispectral index (BIS) is in the range of 40-60.
  Interventions: Drug: propofol infusion

INTERVENTIONS:
Drug: propofol bolus — Propofol will be added in bolus doses of 0.5mg/kg.
  Arms: Group bolus
Drug: propofol infusion — Propofol will be administered as 10mg/kg/hour infusion.
  Arms: Group infusion

SUMMARY:
In this study; during the oocyte retrieval procedure, it was aimed to compare two different general anesthesia methods, in which propofol was administered as infusion according to the patient's Bispectral index system (BIS) value or in bolus doses according to the patient's clinic.The hypothesis of the study; during the oocyte retrieval process, when propofol is administered as an infusion and accompanied by BIS monitoring, adequate anesthesia level will be achieved with less amount of bolus doses according to the clinical condition of the patient.

DETAILED DESCRIPTION:
130 patients over the age of 18, ASA I-II, who underwent oocyte retrieval for IVF treatment were included in the study. The patients divided into two groups. In induction, 2mg/kg fentanyl, 40mg lidocaine and 2mg/kg propofol administered to all patients. Patients in group 1; propofol added in bolus doses of 0.5mg/kg. Doses determined according to the clinical condition of the patient. Patients in group 2; propofol administered as 10mg/kg/hour infusion. The infusion dose adjusted so that the Bispectral index (BIS) is in the range of 40-60.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* ASA I-II
* Patients who underwent oocyte retrieval for IVF treatment

Exclusion Criteria:

1. The patient does not want to participate
2. ASA > II patients
3. Patients under 18 years of age
4. Patients who are allergic to the drugs used
5. Patients with mental illness
6. Patients with alcohol or substance addiction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2022-05-27 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2022-08-17 (Actual)

PRIMARY OUTCOMES:
Propofol | up to 1 hour
  The total amount of Propofol (mg) administered during the procedure

SECONDARY OUTCOMES:
Observer's assessment of sedation scale (OSS) | up to 1 hour
  Time to reach 5 on the observer's assessment of sedation scale of the patients
(Post Anesthetic Discharge Scoring System) PADSS | up to 6 hour
  Time of patients to reach PADSS ≥ 9 (Min:0 and Max: 10) PADSS ≥ 9 is suitable for discharge of the patient
(Satisfaction of patients) STF 1 | up to 6 hour
  Patient satisfaction (The scale is in the range of 1-4. 1: the best)
(Satisfaction of gynecologist) STF 2 | up to 1 hour
  Satisfaction of the doctor performing the procedure(The scale is in the range of 1-4. 1: the best)

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi Bilgen, Study Chair — Acibadem University, Acibadem Kozyatagi Hastanesi
Locations (1):
- Acibadem Kozyatagi Hastanesi, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Bilgen S, Erdogan D, Okten SB. Infusion of propofol with bispectral index monitoring does not reduce the amount of propofol used during transvaginal oocyte retrieval procedure. Sci Rep. 2023 Dec 6;13(1):21561. doi: 10.1038/s41598-023-48611-6. PMID 38057377